CLINICAL TRIAL: NCT06159400
Title: Power-assisted Mobility for Children
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: HS26207 (H2023:321)
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2023-11

CONDITIONS: Power Assisted Device; Children, Only

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this project, we intend to explore the experience of children who use a manual wheelchair (MWC), their parent/guardian, and their prescribing therapist after the child is exposed to a power-assist device (PAD) attached to their MWC as a potential mobility alternative. The specific objectives are 1) to explore the children's experience and impressions of using the PAD; 2) To explore the parent/guardians' perspectives on potential application of the PAD for their child, and 3) To explore occupational/physical therapists' perspectives on potential recommendation of, and training with, a PAD for children.

DETAILED DESCRIPTION:
There are currently no published evidence on the benefits of PADs for children; perceptions of appropriateness among children/parents/clinicians; or information on how PAD introduction and training might be best implemented. Given this paucity of evidence, this study intends to create some foundational knowledge and evidence about PAD use among children.

Research Purpose

In this project, we intend to explore the experience of children who use a MWC, their parent/guardian, and their prescribing therapist after they are exposed to a PAD as a potential mobility alternative. The specific objectives are:

* To explore the children's experience and impressions of using the PAD
* To explore the parent/guardians' perspectives on potential application of the PAD for their child
* To explore occupational/physical therapists' perspectives on potential recommendation of, and training with, a PAD for children We will schedule 2 to 3 sessions, between 30 and 60 minutes long, where the child will have an opportunity to try a PAD with their MWC. The sessions will be held at the Rehabilitation Centre for Children (RCC). We will attach a PAD to the child's MWC using a small bracket on the crossbar of the frame; no change or modification to the MWC is required. A physical or occupational therapist will lead the sessions; they will begin with an explanation and introduction to the PAD and then allow the child to practice using the PAD, providing instruction and ensuring safe operation. The sessions will be video recorded so we can review the sessions later when we are analyzing the interview responses; once the study is complete the video recordings will be destroyed.

After the last session, the parent and child will each be asked to participate in a semi-structured interview. The interviews will last about 30 minutes. We anticipate the interviews will be conducted in a private space at RCC immediately following the last session; however, we can also conduct the interviews at a later time and in a location convenient to you (e.g., at your home; a community location; online).

At the interview, parents will be asked about your perspective on your child's experience with using a PAD on their MWC. Parents will be asked questions about the training process and the potential benefits and drawbacks of using and learning to use a PAD. Sample questions include: Tell me about your child's use of a wheelchair; Tell me what you think of the PAD; Do you think you would want your child to use a PAD? The child will also be interviewed and parents can be present at the interview session with the child if they choose. Sample questions include: Tell me what you think of the PAD; How difficult was it to get the hang of the PAD; Would you want to use a PAD.

ELIGIBILITY:
Inclusion Criteria:

* Children (>18 years) among current Rehabilitation Centre for Children clients who use a manual wheelchair
* parents express a willingness or interest to pursue power assisted device use for their child

Exclusion Criteria:

* have insufficient motor, cognitive and development skills to learn to use a power assisted device

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who are current clients at the Rehabilitation Centre for Children
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Child's experience | The semi-structured interview will be conducted after the final (3rd) session of the child being exposed to the power-assisted device.Interviews will last approximately 30 minutes each.
  A semi-structured interview will be used to gain insight into children's experience using a power-assisted device. After a brief introduction, the child will be asked about their own wheelchair (how long they have used it, how often they use it, what do they do with their wheelchair, do they find it difficult or easy, any challenges). They will then be asked about the power assisted device (what did you think about it, how difficult was it to use, did your therapist do anything to help you with the power assisted device, did you get used to using it, what did you like most, what did you like least). They will then be asked if they would want a power assisted device if it was possible to get one. The interview will then be concluded.
Parent/Guardian's experience | The semi-structured interview will be conducted after the final (3rd) session of the child being exposed to the power-assisted device.Interviews will last approximately 30 minutes each.
  A semi-structured interview will be used to gain insight into parent or guardian's experience with their child using a power-assisted device (PAD). After a brief introduction, the parent/guardian will be asked to tell the interviewers about their child's use of a manual wheelchair (MWC) (how long they have used it, how much time do they use their MWC for mobility, difficulties or challenges with the MWC). They will then be asked about the use of the PAD (what did you think the first time you saw it, how do you think your child found using the PAD the first time and did this change, do you think it was any different than their MWC, how difficult do you think it was for your child to learn to use the PAD, how confident would you be with your child's use of the PAD now, what impact did the PAD have on your child's confidence). They would then be asked if they could, hypothetically, get a PAD for their child, if they would want one. The interview will then be concluded.
Therapist's experience | The semi-structured interview will be conducted after the final (3rd) session of the child being exposed to the power-assisted device. Interviews will last approximately 30 minutes each.
  A semi-structured interview will be used to gain insight into therapist's experience with the child using a power-assisted device (PAD). After a short introduction, the therapist will be asked to tell the interviewer about their pervious experience using a PAD (how familiar they are and how easy it was to learn). They will then be asked how easy (or difficult) they found teaching a child to use the PAD (what made teaching difficult, what concerns did you have about a child using a PAD, what activities do you think are most important to address in training a child to use a PAD, was there enough time (2 or 3 sessions) to get a sense of whether a PAD might be appropriate (safe/competent) for a child). The therapist will then be asked what potential applications do they see for this child using a PAD? The therapist will be asked if they see a potential application for using PAD with other children. The interview will then be concluded.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Giesbrecht, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Kenyon LK, Blank K, Meengs J, Schultz AM. "Make it fun": a qualitative study exploring key aspects of power mobility interventions for children. Disabil Rehabil Assist Technol. 2023 Apr;18(3):304-312. doi: 10.1080/17483107.2020.1849431. Epub 2020 Dec 1. PMID 33259252
- [Background] Ross T, Buliung R. A systematic review of disability's treatment in the active school travel and children's independent mobility literatures. Transport reviews. 2018;38(3):349-371.